CLINICAL TRIAL: NCT04929301
Title: Feasibility and Acceptability of Antenatal Breast Milk Expression-a Pilot Randomized Trial in Nulliparous Pregnant People
Brief Title: Antenatal Milk Expression in Nulliparous Pregnant People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Nurses Foundation (Other)
Responsible Party: Principal Investigator, Jill R. Demirci, PhD, RN, IBCLC, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20040354
Record Dates: First submitted 2021-05-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Pregnancy Related; Breast Feeding; Milk Expression, Breast
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AME Hand-Expression (Experimental): Participants in the antenatal milk expression (AME) group will learn hand-expression from a certified lactation consultant beginning at 37 weeks of pregnancy. At the same visit, the PI or RA will also provide oral and written instructions for AME at home, specifically instructing participants to do AME 1-2 times per day for no longer than 10 minutes.
  Interventions: Other: Antenatal milk expression
- Education (Active Comparator): Participants in the education group will receive a weekly educational hand-out on varying breastfeeding topics (e.g., latch).
  Interventions: Other: Education handouts

INTERVENTIONS:
Other: Antenatal milk expression — Hand-expression of breast milk in pregnancy
  Arms: AME Hand-Expression
Other: Education handouts — Educational breastfeeding handouts
  Arms: Education

SUMMARY:
This was a pilot randomized trial to examine the feasibility and preliminary effectiveness of a structured antenatal milk expression (AME) educational intervention on breastfeeding outcomes within a sample of low-risk pregnant individuals without other children. A convenience sample of 45 participants were enrolled and randomized to either the AME intervention or a control group receiving breastfeeding educational handouts. Both groups met with study staff at 37, 38, 39, and 40 weeks gestation to receive assigned intervention. AME participants practiced AME 1-2 times/day and recorded this in a diary. Data were collected from surveys, interviews, and electronic health record to 3-4 months postpartum.

DETAILED DESCRIPTION:
Antenatal milk expression (AME) has emerged as a simple, inexpensive, novel method to increase maternal breastfeeding confidence, avoid early formula use, and increase proportion of mother's own milk (MOM) feeds-potentially leading to greater breastfeeding satisfaction, increased breastfeeding duration and exclusivity, and improved maternal-infant health outcomes. AME capitalizes on the production, and sometimes leaking, of milk-commencing during the second trimester of pregnancy by allowing women to collect and store milk for later use if needed and gain confidence in breastfeeding and their milk-making capabilities. AME may also "prime" the hormonal milk production process to create a larger postpartum milk supply. Pilot studies conducted with diabetic women demonstrate AME's safety, feasibility, and preliminary effectiveness in improving breastfeeding rates. AME has yet to be investigated in non-diabetic populations.

In the current study, investigators trialed our study procedures and milk collection and analysis methods, and examined the preliminary effectiveness of AME on breastfeeding outcomes among pregnant people without other biological children. Forty-five healthy, nulliparous women were enrolled and randomized to either a structured AME educational intervention or usual care/control group at Magee-Womens Hospital midwife practice at their 34-36 week prenatal appointment. The Principal Investigator (PI) or an research assistant (RA) met with all participants weekly from 37 weeks until delivery, during postpartum hospitalization, and at 1-2 weeks and 3-4 months postpartum. During visits, the PI/RA collected questionnaire data on maternal health and delivery, stress, depression, as well as outcomes of perceived milk supply and breastfeeding attitude, satisfaction, confidence, continuation and exclusivity. Those randomized to AME were taught the technique at the 37 week visit by a lactation consultant, with instructions to continue 1-2 times/day at home. AME was practiced and reinforced with the lactation consultant at each subsequent visit. Those in the control group received breastfeeding handouts at each prenatal visit. For those in the AME group, the PI/RA also collected a small milk sample at each prenatal visit, along with a written diary documenting AME at home. The PI/RA collected a milk sample from all participants at postpartum visits; samples are stored at University of Pittsburgh School of Nursing lab for subsequent analyses (TBD). The PI/RA conducted semi-structured interviews at 1-2 weeks postpartum with AME participants about their experiences with the intervention. Summary statistics were then calculated for feasibility and breastfeeding outcome data, with significance tests (ANOVA, chi-square) to determine group differences breastfeeding outcomes as applicable. Interview data were analyzed for major themes to refine the intervention for a larger trial.

Data collected in this study were used to revise our AME clinical teaching protocol, AME diaries, and establish standard operating procedures for milk collection and storage for an ongoing, larger randomized trial examining AME's effect on breastfeeding outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant with a single fetus
2. 34-36 6/7 weeks pregnant (calculated from anticipated due date)
3. No other living children and no prior breastfeeding experience
4. Plan to breastfeed exclusively for at least 4 months
5. At least 18 years old
6. Plan to deliver baby at Magee-Womens Hospital of UPMC
7. Healthy (no major medical or pregnancy condition which would constitute a high-risk pregnancy)

Exclusion Criteria:

1. Women with contraindications to breastfeeding, as specified by American Academy of Pediatrics, including HIV+ status, human T-cell lymphotrophic virus, etc. HIV status will be assessed by history (maternal self-report of diagnosis).
2. Conditions known to significantly adversely impact maternal milk supply (e.g., breast hypoplasia, history of breast reduction surgery, as assessed on screening form)
3. Conditions which predispose to preterm labor or otherwise constitute a high-risk pregnancy as outlined by the National Institute of Child Health and Human Development including: breech presentation, vaginal bleeding during second or third pregnancy trimester (more than one episode, not related to possible cervical mechanical trauma from sexual intercourse or cervical exam), diagnosed or suspected developmental abnormalities in the fetus, less than 6 months between last birth and the beginning of current pregnancy, placenta previa, diabetes type I or II or gestational diabetes, preeclampsia (or hypertension with proteinuria), smoking, alcohol use, or illicit drug use during pregnancy, oligohydramnios/polyhydramnios, any previous second or third trimester pregnancy loss/miscarriage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-09 (Actual)

PRIMARY OUTCOMES:
Proportion of individuals randomized | End date for study recruitment (approximately one year after beginning enrollment)
  Number of individuals randomized divided by number of individuals screened
Proportion of participants completing study | End date for study data collection (approximately one year after beginning enrollment)
  Number of participants completing final study survey divided by number enrolled

SECONDARY OUTCOMES:
Breastfeeding confidence | Enrollment, postpartum hospitalization: an average of 1-3 days postpartum, 1-2 weeks postpartum, 3-4 months postpartum
  between group differences in Breastfeeding Self-Efficacy Scale-SF (short form) scores (score range 14-70 with higher scores indicative of higher self-efficacy)
Perceived milk supply (single item) | During postpartum hospitalization: an average of 1-3 days postpartum, 1-2 weeks postpartum, 3-4 months postpartum
  Between group differences in perceived postpartum milk supply assessed as a single investigator-created item asking "Do you feel you make enough breast milk to satisfy your baby?" with answer options of "yes," "no," or "unsure" (no and unsure dichotomized to yes="no PIM" and no/unsure= "PIM")
Perceived milk supply (scale score) | During postpartum hospitalization: an average of 1-3 days postpartum, 1-2 weeks postpartum, 3-4 months postpartum
  Between group differences in perceived postpartum milk supply assessed as a combined score on both the Perceived Infant Breastfeeding Satiety and Maternal-Infant Breastfeeding Satisfaction subscales (10 items total) within the H&H Lactation Scale; possible scores range from 0-70, wherein lower scores represented lower breastfeeding satisfaction and lower confidence that one was making enough milk.
In-hospital formula use | Discharge from birth hospital: an average of 1-3 days postpartum
  Between group differences in any formula feeds during birth hospitalization (yes/no) extracted from electronic health record
Breastfeeding continuation | 1-2 weeks postpartum, 3-4 months postpartum
  Between group differences in any breastmilk feeds (yes/no)
Breastfeeding exclusivity | 1-2 weeks postpartum, 3-4 months postpartum
  Between group differences in only breast milk feeds (100% breast milk-yes/no)
Promoters and barriers to antenatal milk collection and storage | 1-2 weeks postpartum
  Qualitative interviews assessing participant perceptions related to collecting and storing antenatal milk
Proportion of participants completing study visits | Study visits at 37, 38, 39, and 40 weeks of pregnancy
  Number of participants completing each study visit divided by number enrolled
Proportion of participants engaging in AME | End date for participant's pregnancy: an average of 40 gestational weeks with upper range to 42 gestational weeks
  Number of participants engaging in AME during study visits and/or independently as documented in AME diary, divided by number of participants assigned to AME

CONTACTS AND LOCATIONS:
Overall Officials: Jill R Demirci, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Magee Women's Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demirci JR, Glasser M, Himes KP, Sereika SM. Structured antenatal milk expression education for nulliparous pregnant people: results of a pilot, randomized controlled trial in the United States. Int Breastfeed J. 2022 Jul 7;17(1):50. doi: 10.1186/s13006-022-00491-8. PMID 35799299